CLINICAL TRIAL: NCT05664347
Title: Video-based Teach-to-goal Intervention on Inhaler Technique on Adults With Asthma and COPD: a Randomized Controlled Trial
Brief Title: Video-based Teach-to-goal Intervention on Inhaler Technique on Jordanian Adults With Asthma and COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Oriana Awwad, Professor, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 124454
Record Dates: First submitted 2022-09-30; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: COPD; Asthma; Inhaled Steroid Dependent Asthma
Keywords: Video-Based; Teach To Goal Education; Chronic Obstructive Pulmonary Disease; Asthma; Randomized Controlled Trial; Patient Education; Quality of Life; Medication adherence; Inhaler technique
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Medication Adherence

STUDY DESIGN:
Intervention Model Description: Patients diagnosed with asthma or COPD, who were started on any inhaler for a minimum of one month and will continue using them chronically were met in the JUH respiratory clinic and invited to participate.
  Patients at high risk for infection, or those presenting with a very severe clinical presentation were excluded.
  Taking into account the non-invasive nature of the educational intervention, and the need to reduce the risk of spread of COVID19 virus (sharing pens or papers), a verbal consent was obtained.
  Enrolled participants were randomized using simple randomization into two groups; odd numbers for the control group (received a verbal TTG education on their inhaler technique) and even numbers for the intervention group ( received a video based TTG education). The primary and secondary outcomes of the study were inhaler technique mastery, amelioration of disease control, disease related quality of life and medication adherence at follow-up (after 3 months).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Standard verbal teach to goal inhaler technique education
  Interventions: Behavioral: Verbal teach to goal education
- Intervention (Active Comparator): Video based teach to goal inhaler technique education
  Interventions: Behavioral: Video based teach to goal education

INTERVENTIONS:
Behavioral: Verbal teach to goal education — Participants were showed how to use correctly their inhalers and then asked again to show the technique. For each incorrect step, the patients were corrected and asked to repeat the steps until they mastered the technique. This process was repeated a maximum of three times.
  Other Names: verbal TTG
  Arms: Control
Behavioral: Video based teach to goal education — Participants were educated by the a video-based teach to goal method. using a smartphone, an educational video illustrating the correct technique for each of the inhalers used by the patient was displayed. After watching the video, the patients were asked to show again how to use their inhaler and for each wrong step the video was displayed again until mastering the correct technique a maximum of three times. At the end of the interview participants in the intervention group received a copy of the video via WhatsApp and were all invited to watch the video whenever needed.
  Other Names: video-based TTG
  Arms: Intervention

SUMMARY:
This study was an interventional educational study that was intended to find out the effect of a video based inhaler technique education on improving inhaler technique mastery, disease control, medication adherence and patient quality of life in comparison to verbal education among adults with asthma or COPD.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of Asthma or COPD.
* Started on one or more inhaler devices for a minimum of one month.
* Expected to continue using their inhaler devices chronically.

Exclusion Criteria:

* Patients at high risk of infection (immunocompromised).
* Patients presenting with a very severe clinical presentation (severe dyspnoea, confusion due to hypoxemia, the need for continuous oxygen therapy).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2021-02-21 (Actual); Study Completion 2021-02-21 (Actual)

PRIMARY OUTCOMES:
Number of participants with correct Inhaler technique | At base line "first interview"
  The ability of the participants to use their inhaler devices correctly: using standardized checklists
Number of participants with correct Inhaler technique | After three months of intervention "second interview"
  The ability of the participants to use their inhaler devices correctly: using standardized checklists

SECONDARY OUTCOMES:
Number of participants with moderate-high medication adherence | At base line "first interview"
  Adherence to inhaled medications used for the management of Asthma or COPD using morisky-green levien scale (MGLS). This scale is a 4 point previously validated score for the assessment of medication adherence, increase in score from 1 to 4 means better medication adherence. patients with a MGLS of 1 were considered to have low medication adherence while those with a score that is equal or higher than 2 were considered to have moderate-high level of adherence.
Number of participants with moderate-high medication adherence | After Three months of intervention "second interview"
  Adherence to inhaled medications used for the management of Asthma or COPD using morisky-green levien scale (MGLS). This scale is a 4 point previously validated score for the assessment of medication adherence, increase in score from 1 to 4 means better medication adherence. patients with a MGLS of 1 were considered to have low medication adherence while those with a score that is equal or higher than 2 were considered to have moderate-high level of adherence.
Number of asthmatic patients with well-controlled Disease | At base line "first interview"
  Assessment of symptom frequency and severity using the Asthma control test (ACT). a scale of 25 points, the minimum score is 5 points which indicates the worst symptom control while the maximum score "best disease control" is indicated by the score of 25.
  Patients with a score of 5-19 were considered having uncontrolled asthma while those with a score of 20-25 had a well controlled asthma.
Number of asthmatic patients with well-controlled Disease | After Three months of intervention "second interview"
  Assessment of symptom frequency and severity using the Asthma control test (ACT). a scale of 25 points, the minimum score is 5 points which indicates the worst symptom control while the maximum score "best disease control" is indicated by the score of 25.
  Patients with a score of 5-19 were considered having uncontrolled asthma while those with a score of 20-25 had a well controlled asthma.
Number of COPD patients with well-controlled Disease | At base line "first interview"
  Assessment of symptom frequency and severity using the COPD assessment test. a scale of 40 points; disease control is considered better as the score decreases. participants with scores of 0-9 were considered having less symptoms "well controlled COPD" while those with a score between 10-40 were considered having more symptoms "less controlled COPD".
Number of COPD patients with well-controlled Disease | After Three months of intervention "second interview"
  Assessment of symptom frequency and severity using the COPD assessment test. a scale of 40 points; disease control is considered better as the score decreases. participants with scores of 0-9 were considered having less symptoms "well controlled COPD" while those with a score between 10-40 were considered having more symptoms "less controlled COPD".
Asthma related quality of life | At base line "first interview"
  Assessment of asthmatic patients quality of life using the mini asthma quality of life questionnaire (mini-AQLQ). A 15 questions scale with a score of 1-7 for each question. average score was calculated to give a result between 1-7. as the average score increased from 1-7 the disease related quality of life was considered better;
  1. total impairment
  2. highly impaired
  3. very impaired
  4. moderately impaired
  5. somehow impaired
  6. little impairment
  7. no impairment.
Asthma related quality of life | After Three months of intervention "second interview"
  Assessment of asthmatic patients quality of life using the mini asthma quality of life questionnaire (mini-AQLQ). A 15 questions scale with a score of 1-7 for each question. average score was calculated to give a result between 1-7. as the average score increased from 1-7 the disease related quality of life was considered better;
  1. total impairment
  2. highly impaired
  3. very impaired
  4. moderately impaired
  5. somehow impaired
  6. little impairment
  7. no impairment.
COPD related quality of life | At base line "first interview"
  Assessment of COPD patients quality of life using the St.George respiratory questionnaire.
  a 50-item validated tool. Each question had a specific weight assigned by the developer and the SGRQ scores are calculated using an automated application that was also designed and afforded by the questionnaire developer.
  The automated application can thus produce four final results; a total score that represents the total burden of COPD on the patient's quality of life, a 'symptom' score, an 'activity limitation' score and an 'impact' score.
  The total SGRQ score and the score for each of the three domains can range from 0 to 100, where an increase in the score indicates more impairment exerted by the disease on the patient's QoL.
COPD related quality of life | After Three months of intervention "second interview"
  Assessment of COPD patients quality of life using the St.George respiratory questionnaire.
  a 50-item validated tool. Each question had a specific weight assigned by the developer and the SGRQ scores are calculated using an automated application that was also designed and afforded by the questionnaire developer.
  The automated application can thus produce four final results; a total score that represents the total burden of COPD on the patient's quality of life, a 'symptom' score, an 'activity limitation' score and an 'impact' score.
  The total SGRQ score and the score for each of the three domains can range from 0 to 100, where an increase in the score indicates more impairment exerted by the disease on the patient's QoL.

CONTACTS AND LOCATIONS:
Locations (1):
- Jordan University Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] G.I.f.C.O.L.D. (GOLD), Global Strategy for the Diagnosis, Managment, and Prevention of Chronic Obstructive Pulmonary Disease, 2020. https://goldcopd.org/gold-reports/. (Accessed November 11, 2019.
- [Background] G.I.f.A. (GINA), Global Strategy for Ashtma Managment and Prevention, 2021. https://ginasthma.org/gina-reports/. (Accessed June 15, 2021.
- [Background] W.H.O. WHO, Chronic Obstructive Pulmonary Disease (COPD) 2017. https://www.who.int/news-room/fact-sheets/detail/chronic-obstructive-pulmonary-disease-(copd). (Accessed January, 22 2020.
- [Background] W.H.O. WHO, Asthma, 2020. https://www.who.int/news-room/q-a-detail/asthma. (Accessed May, 24 2020.
- [Background] European Respiratory Society, The Global Impact of Respiratory Disease, Sheffield, 2017.
- [Background] The global asthma report (GAR), The Burden of Asthma, 2018. http://www.globalasthmareport.org/burden/mortality.php. (Accessed February, 18 2020.
- [Background] Lokke A, Lange P, Lykkegaard J, Ibsen R, Andersson M, de Fine Licht S, Hilberg O. Economic Burden of COPD by Disease Severity - A Nationwide Cohort Study in Denmark. Int J Chron Obstruct Pulmon Dis. 2021 Mar 10;16:603-613. doi: 10.2147/COPD.S295388. eCollection 2021. PMID 33731990
- [Background] C.f.D.C.a.P. CDC, Chronic obstructive pulmonary disease (COPD), 2021. https://www.cdc.gov/copd/infographics/copd-costs.html. (Accessed Jan, 11 2021 2021).
- [Background] Abu-Ekteish F, Otoom S, Shehabi I. Prevalence of asthma in Jordan: comparison between Bedouins and urban schoolchildren using the International Study of Asthma and Allergies in Childhood phase III protocol. Allergy Asthma Proc. 2009 Mar-Apr;30(2):181-5. doi: 10.2500/aap.2009.30.3208. PMID 19463207
- [Background] Khassawneh BY, Samrah SM, Jarrah MI, Ibdah RK, Ibnian AM, Al-Mistarehi AW, Zghayer AA, Abuqudairi SI, Khader YS. Prevalence of undiagnosed COPD in male patients with coronary artery disease: a cross-sectional study in Jordan. Int J Chron Obstruct Pulmon Dis. 2018 Sep 5;13:2759-2766. doi: 10.2147/COPD.S172679. eCollection 2018. PMID 30233166
- [Background] Lavorini F, Fontana GA, Usmani OS. New inhaler devices - the good, the bad and the ugly. Respiration. 2014;88(1):3-15. doi: 10.1159/000363390. Epub 2014 May 27. PMID 24902629
- [Background] Melani AS, Bonavia M, Cilenti V, Cinti C, Lodi M, Martucci P, Serra M, Scichilone N, Sestini P, Aliani M, Neri M; Gruppo Educazionale Associazione Italiana Pneumologi Ospedalieri. Inhaler mishandling remains common in real life and is associated with reduced disease control. Respir Med. 2011 Jun;105(6):930-8. doi: 10.1016/j.rmed.2011.01.005. Epub 2011 Mar 2. PMID 21367593
- [Background] Basheti IA, Obeidat NM, Ammari WG, Reddel HK. Associations between inhaler technique and asthma control among asthma patients using pressurised MDIs and DPIs. Int J Tuberc Lung Dis. 2016 May;20(5):689-95. doi: 10.5588/ijtld.15.0557. PMID 27084826
- [Background] Duarte-de-Araujo A, Teixeira P, Hespanhol V, Correia-de-Sousa J. COPD: misuse of inhaler devices in clinical practice. Int J Chron Obstruct Pulmon Dis. 2019 May 30;14:1209-1217. doi: 10.2147/COPD.S178040. eCollection 2019. PMID 31213798
- [Background] Basheti IA, Obeidat NM, Reddel HK. Inhaler technique education and asthma control among patients hospitalized for asthma in Jordan. Saudi Pharm J. 2018 Dec;26(8):1127-1136. doi: 10.1016/j.jsps.2018.06.002. Epub 2018 Jul 7. PMID 30532633
- [Background] S.J. Hashmi A, Memon A, Soomro T, Incorrect Inhaler Technique Compromising Quality of Life of Asthmatic Patients, Journal of Medicine 13(1) (2012).
- [Background] Usmani OS, Lavorini F, Marshall J, Dunlop WCN, Heron L, Farrington E, Dekhuijzen R. Critical inhaler errors in asthma and COPD: a systematic review of impact on health outcomes. Respir Res. 2018 Jan 16;19(1):10. doi: 10.1186/s12931-017-0710-y. PMID 29338792
- [Background] Sriram KB, Percival M. Suboptimal inhaler medication adherence and incorrect technique are common among chronic obstructive pulmonary disease patients. Chron Respir Dis. 2016 Feb;13(1):13-22. doi: 10.1177/1479972315606313. Epub 2015 Sep 22. PMID 26396159
- [Background] Khurana AK, Dubey K, Goyal A, Pawar KS, Phulwaria C, Pakhare A. Correcting inhaler technique decreases severity of obstruction and improves quality of life among patients with obstructive airway disease. J Family Med Prim Care. 2019 Jan;8(1):246-250. doi: 10.4103/jfmpc.jfmpc_259_18. PMID 30911514
- [Background] Takemura M, Mitsui K, Itotani R, Ishitoko M, Suzuki S, Matsumoto M, Aihara K, Oguma T, Ueda T, Kagioka H, Fukui M. Relationships between repeated instruction on inhalation therapy, medication adherence, and health status in chronic obstructive pulmonary disease. Int J Chron Obstruct Pulmon Dis. 2011;6:97-104. doi: 10.2147/COPD.S16173. Epub 2011 Jan 20. PMID 21407822
- [Background] Takemura M, Kobayashi M, Kimura K, Mitsui K, Masui H, Koyama M, Itotani R, Ishitoko M, Suzuki S, Aihara K, Matsumoto M, Oguma T, Ueda T, Kagioka H, Fukui M. Repeated instruction on inhalation technique improves adherence to the therapeutic regimen in asthma. J Asthma. 2010 Mar;47(2):202-8. doi: 10.3109/02770900903581692. PMID 20170330
- [Background] Baker DW, DeWalt DA, Schillinger D, Hawk V, Ruo B, Bibbins-Domingo K, Weinberger M, Macabasco-O'Connell A, Pignone M. "Teach to goal": theory and design principles of an intervention to improve heart failure self-management skills of patients with low health literacy. J Health Commun. 2011;16 Suppl 3(Suppl 3):73-88. doi: 10.1080/10810730.2011.604379. PMID 21951244
- [Background] Press VG, Arora VM, Trela KC, Adhikari R, Zadravecz FJ, Liao C, Naureckas E, White SR, Meltzer DO, Krishnan JA. Effectiveness of Interventions to Teach Metered-Dose and Diskus Inhaler Techniques. A Randomized Trial. Ann Am Thorac Soc. 2016 Jun;13(6):816-24. doi: 10.1513/AnnalsATS.201509-603OC. PMID 26998961
- [Background] Basheti IA, Salhi YB, Basheti MM, Hamadi SA, Al-Qerem W. Role of the pharmacist in improving inhaler technique and asthma management in rural areas in Jordan. Clin Pharmacol. 2019 Jul 23;11:103-116. doi: 10.2147/CPAA.S213271. eCollection 2019. PMID 31413644
- [Background] Farwana R, Sheriff A, Manzar H, Farwana M, Yusuf A, Sheriff I. Watch this space: a systematic review of the use of video-based media as a patient education tool in ophthalmology. Eye (Lond). 2020 Sep;34(9):1563-1569. doi: 10.1038/s41433-020-0798-z. Epub 2020 Mar 9. PMID 32152516
- [Background] Correnti CM, Chen SC, Stoff BK. Video-based education about systemic corticosteroids enhances patient knowledge more than verbal education: A randomized controlled trial. Dermatol Online J. 2017 Sep 15;23(9):13030/qt2xh2589c. PMID 29469713
- [Background] Denny MC, Vahidy F, Vu KY, Sharrief AZ, Savitz SI. Video-based educational intervention associated with improved stroke literacy, self-efficacy, and patient satisfaction. PLoS One. 2017 Mar 23;12(3):e0171952. doi: 10.1371/journal.pone.0171952. eCollection 2017. PMID 28333925
- [Background] Lirsac B, Braunstein G. [Randomized evaluation of two teaching methods using aerosol dosers]. Rev Mal Respir. 1991;8(6):559-65. French. PMID 1685595
- [Background] van der Palen J, Klein JJ, Kerkhoff AH, van Herwaarden CL, Seydel ER. Evaluation of the long-term effectiveness of three instruction modes for inhaling medicines. Patient Educ Couns. 1997 Dec;32(1 Suppl):S87-95. doi: 10.1016/s0738-3991(97)00100-6. PMID 9516764
- [Background] Shah RF, Gupta RM. Video instruction is more effective than written instruction in improving inhaler technique. Pulm Pharmacol Ther. 2017 Oct;46:16-19. doi: 10.1016/j.pupt.2017.08.005. Epub 2017 Aug 7. PMID 28797611
- [Background] Windisch W, Schwarz SB, Magnet FS, Dreher M, Schmoor C, Storre JH, Knipel V. Using web-based videos to improve inhalation technique in COPD patients requiring hospitalization: A randomized controlled trial. PLoS One. 2018 Oct 16;13(10):e0201188. doi: 10.1371/journal.pone.0201188. eCollection 2018. PMID 30325931
- [Background] Press VG, Kelly CA, Kim JJ, White SR, Meltzer DO, Arora VM. Virtual Teach-To-Goal Adaptive Learning of Inhaler Technique for Inpatients with Asthma or COPD. J Allergy Clin Immunol Pract. 2017 Jul-Aug;5(4):1032-1039.e1. doi: 10.1016/j.jaip.2016.11.018. Epub 2017 Jan 5. PMID 28065689
- [Background] Basheti IA, Obeidat NM, Reddel HK. Effect of novel inhaler technique reminder labels on the retention of inhaler technique skills in asthma: a single-blind randomized controlled trial. NPJ Prim Care Respir Med. 2017 Feb 9;27(1):9. doi: 10.1038/s41533-017-0011-4. PMID 28184045
- [Background] Almomani BA, Mokhemer E, Al-Sawalha NA, Momany SM. A novel approach of using educational pharmaceutical pictogram for improving inhaler techniques in patients with asthma. Respir Med. 2018 Oct;143:103-108. doi: 10.1016/j.rmed.2018.09.004. Epub 2018 Sep 6. PMID 30261980
- [Background] Department of health UAE, Asthma control test for 12 years or older, 2019. https://www.doh.gov.ae/programs-initiatives/chronic-respiratory-diseases-awareness-program. (Accessed 2021, April 18.
- [Background] Lababidi H, Hijaoui A, Zarzour M. Validation of the Arabic version of the asthma control test. Ann Thorac Med. 2008 Apr;3(2):44-7. doi: 10.4103/1817-1737.39635. PMID 19561904
- [Background] Al-Moamary MS, Al-Hajjaj MS, Tamim HM, Al-Ghobain MO, Al-Qahtani HA, Al-Kassimi FA. The reliability of an Arabic translation of the chronic obstructive pulmonary disease assessment test. Saudi Med J. 2011 Oct;32(10):1028-33. PMID 22008922
- [Background] Juniper EF, Guyatt GH, Cox FM, Ferrie PJ, King DR. Development and validation of the Mini Asthma Quality of Life Questionnaire. Eur Respir J. 1999 Jul;14(1):32-8. doi: 10.1034/j.1399-3003.1999.14a08.x. PMID 10489826
- [Background] S.G.u.o. London, St George's Respiratory Questionnaire (SGRQ), 2021. https://www.sgul.ac.uk/about/our-institutes/infection-and-immunity/research-themes/research-centres/health-status. (Accessed April, 7 2021).
- [Background] Morisky DE, Green LW, Levine DM. Concurrent and predictive validity of a self-reported measure of medication adherence. Med Care. 1986 Jan;24(1):67-74. doi: 10.1097/00005650-198601000-00007. PMID 3945130
- [Background] The Deutsche Atemwegsliga (German Airway League), Breezhaler (Mono) الاستنشاق بجهاز بريزهيلر, 2016.
- [Background] ClinCalc, Sample size calculator. https://clincalc.com/stats/samplesize.aspx. (Accessed March, 5 2020.
- [Background] Al Omari M, Khassawneh BY, Khader Y, Dauod AS, Bergus G. Prevalence of chronic obstructive pulmonary disease among adult male cigarettes smokers: a community-based study in Jordan. Int J Chron Obstruct Pulmon Dis. 2014 Jul 17;9:753-8. doi: 10.2147/COPD.S62898. eCollection 2014. PMID 25092972
- [Background] Mohamed Hoesein FA, Zanen P, Lammers JW. Lower limit of normal or FEV1/FVC < 0.70 in diagnosing COPD: an evidence-based review. Respir Med. 2011 Jun;105(6):907-15. doi: 10.1016/j.rmed.2011.01.008. Epub 2011 Feb 5. PMID 21295958
- [Background] Normansell R, Kew KM, Mathioudakis AG. Interventions to improve inhaler technique for people with asthma. Cochrane Database Syst Rev. 2017 Mar 13;3(3):CD012286. doi: 10.1002/14651858.CD012286.pub2. PMID 28288272
- [Background] Jahedi L, Downie SR, Saini B, Chan HK, Bosnic-Anticevich S. Inhaler Technique in Asthma: How Does It Relate to Patients' Preferences and Attitudes Toward Their Inhalers? J Aerosol Med Pulm Drug Deliv. 2017 Feb;30(1):42-52. doi: 10.1089/jamp.2016.1287. Epub 2016 Sep 27. PMID 27676193
- [Background] van der Palen J, Klein JJ, van Herwaarden CL, Zielhuis GA, Seydel ER. Multiple inhalers confuse asthma patients. Eur Respir J. 1999 Nov;14(5):1034-7. doi: 10.1183/09031936.99.14510349. PMID 10596686
- [Background] Press VG, Arora VM, Shah LM, Lewis SL, Ivy K, Charbeneau J, Badlani S, Nareckas E, Mazurek A, Krishnan JA. Misuse of respiratory inhalers in hospitalized patients with asthma or COPD. J Gen Intern Med. 2011 Jun;26(6):635-42. doi: 10.1007/s11606-010-1624-2. Epub 2011 Jan 20. PMID 21249463
- [Background] Press VG, Arora VM, Shah LM, Lewis SL, Charbeneau J, Naureckas ET, Krishnan JA. Teaching the use of respiratory inhalers to hospitalized patients with asthma or COPD: a randomized trial. J Gen Intern Med. 2012 Oct;27(10):1317-25. doi: 10.1007/s11606-012-2090-9. Epub 2012 May 17. PMID 22592354
- [Background] Bosnic-Anticevich SZ, Sinha H, So S, Reddel HK. Metered-dose inhaler technique: the effect of two educational interventions delivered in community pharmacy over time. J Asthma. 2010 Apr;47(3):251-6. doi: 10.3109/02770900903580843. PMID 20394511
- [Background] Alzayer R, Chaar B, Basheti I, Saini B. Asthma management experiences of Australians who are native Arabic speakers. J Asthma. 2018 Jul;55(7):801-810. doi: 10.1080/02770903.2017.1362702. Epub 2017 Oct 4. PMID 28800268
- [Background] Ovchinikova L, Smith L, Bosnic-Anticevich S. Inhaler technique maintenance: gaining an understanding from the patient's perspective. J Asthma. 2011 Aug;48(6):616-24. doi: 10.3109/02770903.2011.580032. Epub 2011 May 31. PMID 21623690
- [Background] Pothirat C, Chaiwong W, Phetsuk N, Pisalthanapuna S, Chetsadaphan N, Choomuang W. Evaluating inhaler use technique in COPD patients. Int J Chron Obstruct Pulmon Dis. 2015 Jul 8;10:1291-8. doi: 10.2147/COPD.S85681. eCollection 2015. PMID 26185435
- [Background] Fink JB, Rubin BK. Problems with inhaler use: a call for improved clinician and patient education. Respir Care. 2005 Oct;50(10):1360-74; discussion 1374-5. PMID 16185371
- [Background] Karle E, Patel TP, Zweig J, Krvavac A. Understanding the Knowledge Gap and Assessing Comfort Level among Healthcare Professionals Who Provide Inhaler Education. COPD. 2020 Apr;17(2):197-204. doi: 10.1080/15412555.2020.1746251. Epub 2020 Apr 1. PMID 32237908
- [Background] Nimmo CJ, Chen DN, Martinusen SM, Ustad TL, Ostrow DN. Assessment of patient acceptance and inhalation technique of a pressurized aerosol inhaler and two breath-actuated devices. Ann Pharmacother. 1993 Jul-Aug;27(7-8):922-7. doi: 10.1177/106002809302700721. PMID 8364279
- [Background] Baker DW, Dewalt DA, Schillinger D, Hawk V, Ruo B, Bibbins-Domingo K, Weinberger M, Macabasco-O'Connell A, Grady KL, Holmes GM, Erman B, Broucksou KA, Pignone M. The effect of progressive, reinforcing telephone education and counseling versus brief educational intervention on knowledge, self-care behaviors and heart failure symptoms. J Card Fail. 2011 Oct;17(10):789-96. doi: 10.1016/j.cardfail.2011.06.374. Epub 2011 Jul 23. PMID 21962415
- [Background] Basheti IA, Armour CL, Bosnic-Anticevich SZ, Reddel HK. Evaluation of a novel educational strategy, including inhaler-based reminder labels, to improve asthma inhaler technique. Patient Educ Couns. 2008 Jul;72(1):26-33. doi: 10.1016/j.pec.2008.01.014. Epub 2008 Mar 7. PMID 18314294
- [Background] Giraud V, Allaert FA, Roche N. Inhaler technique and asthma: feasability and acceptability of training by pharmacists. Respir Med. 2011 Dec;105(12):1815-22. doi: 10.1016/j.rmed.2011.07.004. Epub 2011 Jul 28. PMID 21802271
- [Background] Levy ML, Hardwell A, McKnight E, Holmes J. Asthma patients' inability to use a pressurised metered-dose inhaler (pMDI) correctly correlates with poor asthma control as defined by the global initiative for asthma (GINA) strategy: a retrospective analysis. Prim Care Respir J. 2013 Dec;22(4):406-11. doi: 10.4104/pcrj.2013.00084. PMID 24042172
- [Background] George M, Bender B. New insights to improve treatment adherence in asthma and COPD. Patient Prefer Adherence. 2019 Jul 31;13:1325-1334. doi: 10.2147/PPA.S209532. eCollection 2019. PMID 31534319
- [Background] Harnett CM, Hunt EB, Bowen BR, O'Connell OJ, Edgeworth DM, Mitchell P, Eustace JA, Henry MT, Kennedy MP, Plant BJ, Murphy DM. A study to assess inhaler technique and its potential impact on asthma control in patients attending an asthma clinic. J Asthma. 2014 May;51(4):440-5. doi: 10.3109/02770903.2013.876650. Epub 2014 Jan 24. PMID 24393080
- [Background] Souza DS, Noblat Lde A, Santos Pde M. Factors associated with quality of life in patients with severe asthma: the impact of pharmacotherapy. J Bras Pneumol. 2015 Nov-Dec;41(6):496-501. doi: 10.1590/S1806-37562015000004545. PMID 26785957
- [Background] Almomani BA, Al-Sawalha NA, Samrah SM, Gamble JM, Al Momani MA. Asthma insights from Jordan: cross-sectional observational study. J Asthma. 2016;53(4):349-55. doi: 10.3109/02770903.2015.1121493. Epub 2016 Jan 22. PMID 26666170
- [Background] Miravitlles M, Molina J, Naberan K, Cots JM, Ros F, Llor C; EVOCA study. Factors determining the quality of life of patients with COPD in primary care. Ther Adv Respir Dis. 2007 Dec;1(2):85-92. doi: 10.1177/1753465807086097. PMID 19124350
- [Background] Schlecht NF, Schwartzman K, Bourbeau J. Dyspnea as clinical indicator in patients with chronic obstructive pulmonary disease. Chron Respir Dis. 2005;2(4):183-91. doi: 10.1191/1479972305cd079oa. PMID 16541601
- [Background] Braido F, Chrystyn H, Baiardini I, Bosnic-Anticevich S, van der Molen T, Dandurand RJ, Chisholm A, Carter V, Price D; Respiratory Effectiveness Group. "Trying, But Failing" - The Role of Inhaler Technique and Mode of Delivery in Respiratory Medication Adherence. J Allergy Clin Immunol Pract. 2016 Sep-Oct;4(5):823-32. doi: 10.1016/j.jaip.2016.03.002. PMID 27587316
- [Background] Vrijens B, Dima AL, Van Ganse E, van Boven JF, Eakin MN, Foster JM, de Bruin M, Chisholm A, Price D. What We Mean When We Talk About Adherence in Respiratory Medicine. J Allergy Clin Immunol Pract. 2016 Sep-Oct;4(5):802-12. doi: 10.1016/j.jaip.2016.05.019. PMID 27587314
- [Derived] Al-Kharouf MS, Abdeljalil MH, Obeidat NM, Oweidat KA, Awwad O. Video-based teach-to-goal intervention on inhaler technique on adults with asthma and COPD: A randomized controlled trial. PLoS One. 2023 Jun 9;18(6):e0286870. doi: 10.1371/journal.pone.0286870. eCollection 2023. PMID 37294823